CLINICAL TRIAL: NCT00283530
Title: Identification of Tumor Phenotypes and Correlation to Clinical Outcomes in Patients Diagnosed With Cancer
Brief Title: Tumor Phenotypes and Correlation to Clinical Outcomes in Cancer
Status: Terminated | Type: Observational
Why Stopped: The PI is no longer with Kentuckiana Cancer Institute. All current subjects completed. No further subjects will be enrolled. Terminated with IRB.
Sponsor: Kentuckiana Cancer Institute (Other)
Other Study IDs: 1050203; CPTAIV-0020-385
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Cancer
Keywords: Cancer; Cancer receiving chemotherapy; Tumor biopsy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Tumor biopsy

SUMMARY:
The purpose of this study is to identify the genetic makeup of cancers, the cancer response, and the correlation of the cancer response to standardized regimens of cancer treatment.

DETAILED DESCRIPTION:
To identify the genetic makeup of cancers, the cancer response, and the correlation of the cancer response to standardized regimens of cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer receiving chemotherapy
* Have had or will have tissue and/or blood samples collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer subjects who have or will have tissue and or blood collected.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2003-05; Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D. Glisson, MD, Study Director — Kentuckiana Cancer Institute
Locations (1):
- Kentuckiana Cancer Institute, Louisville, Kentucky, United States